CLINICAL TRIAL: NCT02056158
Title: HIV+ Alveolar Macrophage Oxidant-mediated Apoptosis of Pulmonary Endothelium
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1307014135; U01HL121828 (NIH)
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: HIV; COPD; Emphysema; Smoking
Keywords: HIV; COPD; Emphysema; Smoking
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples and biopsies from the lower respiratory tract.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- HIV Negative Early COPD Smokers: HIV Negative Early COPD Smokers
- HIV Negative COPD Smokers: HIV Negative COPD Smokers
- HIV Negative Nonsmokers: HIV Negative Nonsmokers
- HIV Negative Smokers: HIV Negative Smokers
- HIV Positive Smokers: HIV Positive Smokers
- HIV Positive Nonsmokers: HIV Positive Nonsmokers
- HIV Positive COPD Smokers: HIV Positive COPD Smokers
- HIV Positive Early COPD Smokers: HIV Positive Early COPD Smokers

SUMMARY:
In HIV+ cigarette smokers, with no prior history of pulmonary infections, emphysema is often developed at an earlier age and is a significant cause of morbidity despite treatment with antiretroviral drugs. Preliminary data gathered from HIV+ individuals that smoke cigarettes strongly support the hypothesis that the combination of HIV infection and smoking creates increased stress in the lower respiratory tract. To examine the underlying factors that contribute to the accelerated development of emphysema in this cohort, samples from the lower respiratory tract will be provided by HIV+ and HIV- subjects. The samples collected will serve as biomarkers for assessing the onset of emphysema.

DETAILED DESCRIPTION:
The purpose of this study is to analyze biologic samples from the blood, airways and/or urine of HIV- and HIV+ smokers and non-smokers to better understand the etiology and pathogenesis of emphysema in association with HIV infection. The underlying hypothesis is that the combination of HIV infection and smoking creates chronic oxidant stress in the lower respiratory tract that promotes cellular loss and contributes to the progressive development of emphysema. Preliminary data strongly supports our hypothesis that the accelerated development of emphysema among HIV+ smokers is due in part to the interaction of HIV directly on the macrophage found in the pulmonary alveolus. The interaction causes a release of exaggerated amounts of oxidants in the lower respiratory tract and leads to increased levels of oxidized metabolites. HIV+ individuals with emphysema have high plasma levels of apoptotic pulmonary capillary-derived micro particles that contain oxidized metabolites. The increased release of micro particles is characteristic of an apoptotic process.

We will study this hypothesis by sampling HIV+ and HIV- subjects alveolar macrophages (AM), which are found on the epithelial surface of the lung, and epithelial lining fluid (ELF) found in the lower respiratory tract. We will also assess plasma pulmonary capillary-derived endothelial microparticles (EMPs) as a biomarker for pulmonary apoptosis. Using newly developed mass spectrometry methodologies, we will quantify the oxidant stress of AM, ELF and plasma EMPs, and identify specific oxidized metabolites within each of these compartments. Finally, we will examine the interaction in vitro to tease apart the contribution of each component (AM, ELF, and plasma EMPs) of the interaction.

To assess this concept, the following aims will be addressed:

Specific Aim 1 (n=160). To explore the extent of the oxidant stress in the lower respiratory tract in association with HIV infection and smoking.

Specific Aim 2 (n=160). To evaluate plasma levels of capillary apoptosis and oxidation state of HIV+ nonsmokers and smokers.

Specific Aim 3 (n=160). To examine the interaction of pulmonary capillary endothelium and various oxidant effector components to identify oxidant-vulnerable pathways relevant to the development of new treatment therapies.

ELIGIBILITY:
Inclusion Criteria:

HEALTHY VOLUNTEER RESEARCH SUBJECTS

* All study subjects should be able to provide informed consent
* Males or females ages 18 years and older
* Must provide HIV informed consent

VOLUNTEER RESEARCH SUBJECTS WITH LUNG DISEASE

* Must provide informed consent
* Males and females age 18 years and older
* Lung disease proven by at least one of the following: symptoms consistent with pulmonary disease; (2) chest X-rays consistent with lung disease; (3) pulmonary function tests consistent with lung disease; (4) lung biopsy consistent with lung disease; (5) family history of lung disease; and/or (6) diseases of organs with known association with lung disease
* Must provide HIV informed consent

Exclusion Criteria:

HEALTHY VOLUNTEER RESEARCH SUBJECTS

* Individuals not deemed in good overall health by the investigator will not be accepted into the study.
* Habitual use of drugs and/or alcohol within the past six months (Acceptable: - Marijuana one time in three months; average of two alcoholic beverages per day; drug and/or alcohol abuse is defined as per the DSM-IV Substance Abuse Criteria).
* Individuals with history of chronic lung disease, including asthma or with recurrent or recent (within three months) acute pulmonary disease will not be accepted into the study.
* Individuals with allergies to atropine or any local anesthetic will not be accepted into the study.
* Individuals with allergies to pilocarpine, isoproterenol, terbutaline, atropine or aminophylline will not be accepted into the study.
* Females who are pregnant or nursing will not be accepted into the study

VOLUNTEER RESEARCH SUBJECTS WITH LUNG DISEASE

* Any history of allergies to xylocaine, lidocaine, versed, valium, atropine, pilocarpine, isoproterenol, terbutaline, aminophylline, or any local anesthetic will not be included in the study.
* Habitual use of drugs and/or alcohol within the past six months (Acceptable: Marijuana one time in three months; average of two alcoholic beverages per day; drug and/or alcohol abuse is defined as per the DSM-IV Substance Abuse Criteria)
* Females who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: New York Metropolitan area residents
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-01-13 (Actual); Primary Completion 2015-10-05 (Actual); Study Completion 2015-10-23 (Actual)

PRIMARY OUTCOMES:
Changes in oxidant stress in the lower respiratory tract in association with HIV infection and smoking | One year
  Using samples obtained from subjects the extent and nature of the HIV/smoking-induced oxidant burden of the lower respiratory tract will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Department of Genetic Medicne, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided